CLINICAL TRIAL: NCT01922700
Title: Pepper Gas Exposure Study
Brief Title: Effects of Pepper Gas Exposure in Non-combatant Bystanders.
Status: Completed | Type: Observational
Sponsor: Sheri Kashmir Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Parvaiz A Koul, Professor & Head, Internal & Pulmonary Medicine, Sheri Kashmir Institute of Medical Sciences
Other Study IDs: PEPPER01
Record Dates: First submitted 2013-08-08; First posted 2013-08-14 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Cough; Irritation in Throat; Irritation in Skin; Lacrimation
Keywords: Pepper spray; bronchospasm; lacrimation
MeSH Terms: conditions — Cough; Lacerations; Bronchial Spasm

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Pepper sprays and pepper gas grenades are used by riot police at various places in the world for crowd control. Data about the acute effects based on human studies is extremely scarce. Kashmir valley in the northern Indian state of Jammu & Kashmir has witnessed political turmoil for the past 22 years and incidents of stone pelting are common wherein groups of youth indulge in stone pelting at the security personnel. While there have been previous episodes of fatalities associated with incidents of firing by the security personnel; non lethal methods are adopted routinely now. These include lathis, water cannons, tear gas and more recently the pepper gas grenades. The pepper grenades explode in the area and the adverse effects are perceived by the population in the area too who are even sitting in their homes. The study proposes to observe the health effects of the pepper gas exposure in non-combatant civilians.

DETAILED DESCRIPTION:
Eligibility:

History of exposure to a pepper grenade explosion.

Exclusion:

Participation in combat operation/ stone pelting/ demonstration.

ELIGIBILITY:
Inclusion Criteria:

All participants with a history of exposure to pepper gas grenade explosion

Exclusion Criteria:

Combatant role while exposure

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community based non-combatant individuals exposed to pepper gases while being used on combatants.
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Development of cough, irritation in throat, nasal irritation, nasal discharge, wheezing, breathlessness, hemoptysis, chest pain upon exposure or worsening of already existing cough, breathlessness, wheezing of a previous respiratory illness. | 24 hours

SECONDARY OUTCOMES:
Duration of symptoms developed | 10 days

OTHER OUTCOMES:
Development of other non-respiratory symptoms which include (but not limited to) skin irritation, skin rash, lacrimation, visual disturbances, vomiting, any other GI symptom, headache, fever, seizures or any other neurological symptom and their duration | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Parvaiz Koul, MD, FRCP, FACP, Principal Investigator — Professor & Head, Internal & Pulmonary Medicine, SKIMS,Srinagar 190011 , J&K (India)
Locations (1):
- SheriKashmir Institute of Medical Sciences, Srinagar, Jammu and Kashmir, India

REFERENCES:
- [Background] Cil H, Atilgan ZA, Islamoglu Y, Tekbas EO, Dostbil Z. Is the pepper spray a triggering factor in myocardial infarction? A case report. Eur Rev Med Pharmacol Sci. 2012 Mar;16 Suppl 1:73-4. PMID 22582490
- [Result] Holopainen JM, Moilanen JA, Hack T, Tervo TM. Toxic carriers in pepper sprays may cause corneal erosion. Toxicol Appl Pharmacol. 2003 Feb 1;186(3):155-62. doi: 10.1016/s0041-008x(02)00015-7. PMID 12620368
- [Result] Vesaluoma M, Muller L, Gallar J, Lambiase A, Moilanen J, Hack T, Belmonte C, Tervo T. Effects of oleoresin capsicum pepper spray on human corneal morphology and sensitivity. Invest Ophthalmol Vis Sci. 2000 Jul;41(8):2138-47. PMID 10892855